CLINICAL TRIAL: NCT06376383
Title: Tonsillectomy Versus Tonsillotomy in Adults With Obstructive Sleep Apnea; a Randomized Controlled Trial Comparing Postoperative Morbidity
Brief Title: Tonsillectomy vs. Tonsillotomy in Adults With Obstructive Sleep Apnea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TETT-RHG; 110500 (Other: The Central Denmark Region Committees on Health Research Ethics)
Record Dates: First submitted 2024-04-09; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea; Tonsillar Hypertrophy
Keywords: Tonsillectomy; Obstructive sleep apnea (OSA); Tonsillotomy; Intracapsular reduction of tonsils; Drug Induced Sedation Endoscopy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Tonsillectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tonsillectomy (Active Comparator): Patients undergo standard removal of subcapsular removal of palatine tonsils
  Interventions: Procedure: Tonsillectomy
- Tonsillotomy (Experimental): Patients undergo intracapsular reduction of palatine tonsils
  Interventions: Procedure: Tonsillotomy

INTERVENTIONS:
Procedure: Tonsillectomy — Standard tonsillectomy
  Other Names: TE
  Arms: Tonsillectomy
Procedure: Tonsillotomy — Tonsillotomy
  Other Names: TT
  Arms: Tonsillotomy

SUMMARY:
The primary purpose of this randomized controlled trial s to investigate whether surgical reduction of palatine tonsils (tonsillotomy) is a superior treatment compared to complete surgical removal of palatine tonsils (tonsillectomy) in adults patients with obstructive sleep apnea and concomitant enlarged tonsils in regards of perioperative and postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Tonsil size 2, 3, or 4 (Friedman tonsil scale)
* Confirmed OSA with sleep analysis not older than a year either CRM or PSG
* ASA 1 or 2
* BMI < 35 kg/m2

Exclusion Criteria:

Children age < 18 years

* Previous pharyngeal surgery such as previous tonsillotomy, tonsillectomy or palatal surgery
* Epileptic disease or severe neurological comorbidity.
* ASA 3, or 4.
* Central sleep apnea
* Previous thrombotic disease.
* Currently treated with sleep medications
* No collapse of oropharyngeal lateral wall during DISE
* Dropout of study, lack of sleep analysis or lack of postoperative DISE.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative hemorrhage | 14 days
  Postoperative hemorrhage event - readmission to the hospital
Postoperative pain | 30 days
  Postoperative pain self-assed daily by using Visual Analoge Scale (VAS) 0 = No pain, 10 = maximal pain.
Recovery time - Sick leave | 30 days
  Sick-leave in days, measured when the patient is at work or back at school, day 0 = surgery day and outcome day is last day of sick-leave
Morbidity | 30 days
  Re-admission at the hospital. Event is registered as null if no re-admission occurs and 1 or 2 etc. if re-admission occurs within first 30 days after surgery

SECONDARY OUTCOMES:
AHI | 180 days
  Apnea Hypopnea Index before and after surgery. Increase in AHI means worsening in apnea hypopnea index. AHI is measured by performing at home type 3 sleep registration
DISE - VOTE | 180 days
  Velum Oropharyngeal Tongue base Epiglottis (VOTE) evaluation. 0 = no collaps
  1. = partial collaps
  2. = complete collaps

REFERENCES:
- [Background] Levy P, Kohler M, McNicholas WT, Barbe F, McEvoy RD, Somers VK, Lavie L, Pepin JL. Obstructive sleep apnoea syndrome. Nat Rev Dis Primers. 2015 Jun 25;1:15015. doi: 10.1038/nrdp.2015.15. PMID 27188535
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Fietze I, Laharnar N, Obst A, Ewert R, Felix SB, Garcia C, Glaser S, Glos M, Schmidt CO, Stubbe B, Volzke H, Zimmermann S, Penzel T. Prevalence and association analysis of obstructive sleep apnea with gender and age differences - Results of SHIP-Trend. J Sleep Res. 2019 Oct;28(5):e12770. doi: 10.1111/jsr.12770. Epub 2018 Oct 1. PMID 30272383
- [Background] Drager LF, McEvoy RD, Barbe F, Lorenzi-Filho G, Redline S; INCOSACT Initiative (International Collaboration of Sleep Apnea Cardiovascular Trialists). Sleep Apnea and Cardiovascular Disease: Lessons From Recent Trials and Need for Team Science. Circulation. 2017 Nov 7;136(19):1840-1850. doi: 10.1161/CIRCULATIONAHA.117.029400. PMID 29109195
- [Background] Young T, Skatrud J, Peppard PE. Risk factors for obstructive sleep apnea in adults. JAMA. 2004 Apr 28;291(16):2013-6. doi: 10.1001/jama.291.16.2013. No abstract available. PMID 15113821
- [Background] Van Ryswyk E, Anderson CS, Antic NA, Barbe F, Bittencourt L, Freed R, Heeley E, Liu Z, Loffler KA, Lorenzi-Filho G, Luo Y, Margalef MJM, McEvoy RD, Mediano O, Mukherjee S, Ou Q, Woodman R, Zhang X, Chai-Coetzer CL. Predictors of long-term adherence to continuous positive airway pressure in patients with obstructive sleep apnea and cardiovascular disease. Sleep. 2019 Oct 9;42(10):zsz152. doi: 10.1093/sleep/zsz152. PMID 31587046
- [Background] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- [Background] Kezirian EJ, Hohenhorst W, de Vries N. Drug-induced sleep endoscopy: the VOTE classification. Eur Arch Otorhinolaryngol. 2011 Aug;268(8):1233-1236. doi: 10.1007/s00405-011-1633-8. Epub 2011 May 26. PMID 21614467
- [Background] Lechner M, Wilkins D, Kotecha B. A review on drug-induced sedation endoscopy - Technique, grading systems and controversies. Sleep Med Rev. 2018 Oct;41:141-148. doi: 10.1016/j.smrv.2018.02.001. Epub 2018 Feb 24. PMID 29627276
- [Background] MacKay S, Carney AS, Catcheside PG, Chai-Coetzer CL, Chia M, Cistulli PA, Hodge JC, Jones A, Kaambwa B, Lewis R, Ooi EH, Pinczel AJ, McArdle N, Rees G, Singh B, Stow N, Weaver EM, Woodman RJ, Woods CM, Yeo A, McEvoy RD. Effect of Multilevel Upper Airway Surgery vs Medical Management on the Apnea-Hypopnea Index and Patient-Reported Daytime Sleepiness Among Patients With Moderate or Severe Obstructive Sleep Apnea: The SAMS Randomized Clinical Trial. JAMA. 2020 Sep 22;324(12):1168-1179. doi: 10.1001/jama.2020.14265. PMID 32886102
- [Background] Rashwan MS, Montevecchi F, Cammaroto G, Badr El Deen M, Iskander N, El Hennawi D, El Tabbakh M, Meccariello G, Gobbi R, Stomeo F, Vicini C. Evolution of soft palate surgery techniques for obstructive sleep apnea patients: A comparative study for single-level palatal surgeries. Clin Otolaryngol. 2018 Apr;43(2):584-590. doi: 10.1111/coa.13027. Epub 2017 Dec 3. PMID 29106778
- [Background] Camacho M, Li D, Kawai M, Zaghi S, Teixeira J, Senchak AJ, Brietzke SE, Frasier S, Certal V. Tonsillectomy for adult obstructive sleep apnea: A systematic review and meta-analysis. Laryngoscope. 2016 Sep;126(9):2176-86. doi: 10.1002/lary.25931. Epub 2016 Mar 22. PMID 27005314
- [Background] Reckley LK, Fernandez-Salvador C, Camacho M. The effect of tonsillectomy on obstructive sleep apnea: an overview of systematic reviews. Nat Sci Sleep. 2018 Apr 4;10:105-110. doi: 10.2147/NSS.S127816. eCollection 2018. PMID 29670412
- [Background] Sjoblom HM, Nahkuri M, Suomela M, Jero J, Piitulainen JM. Treatment of sleep apnoea with tonsillectomy: a retrospective analysis using long-term follow-up data. Eur Arch Otorhinolaryngol. 2022 Jul;279(7):3727-3732. doi: 10.1007/s00405-022-07350-6. Epub 2022 Mar 25. PMID 35338397
- [Background] Randall DA, Hoffer ME. Complications of tonsillectomy and adenoidectomy. Otolaryngol Head Neck Surg. 1998 Jan;118(1):61-8. doi: 10.1016/S0194-5998(98)70376-6. PMID 9450830
- [Background] Myssiorek D, Alvi A. Post-tonsillectomy hemorrhage: an assessment of risk factors. Int J Pediatr Otorhinolaryngol. 1996 Sep;37(1):35-43. doi: 10.1016/0165-5876(96)01364-x. PMID 8884405
- [Background] Zhang LY, Zhong L, David M, Cervin A. Tonsillectomy or tonsillotomy? A systematic review for paediatric sleep-disordered breathing. Int J Pediatr Otorhinolaryngol. 2017 Dec;103:41-50. doi: 10.1016/j.ijporl.2017.10.008. Epub 2017 Oct 5. PMID 29224763
- [Background] Wang H, Fu Y, Feng Y, Guan J, Yin S. Tonsillectomy versus tonsillotomy for sleep-disordered breathing in children: a meta analysis. PLoS One. 2015 Mar 25;10(3):e0121500. doi: 10.1371/journal.pone.0121500. eCollection 2015. PMID 25807322
- [Background] Acevedo JL, Shah RK, Brietzke SE. Systematic review of complications of tonsillotomy versus tonsillectomy. Otolaryngol Head Neck Surg. 2012 Jun;146(6):871-9. doi: 10.1177/0194599812439017. Epub 2012 Mar 6. PMID 22394550
- [Background] Wong Chung JERE, van Benthem PPG, Blom HM. Tonsillotomy versus tonsillectomy in adults suffering from tonsil-related afflictions: a systematic review. Acta Otolaryngol. 2018 May;138(5):492-501. doi: 10.1080/00016489.2017.1412500. Epub 2017 Dec 15. PMID 29241412